CLINICAL TRIAL: NCT02070731
Title: A Prospective, Randomized Evaluation of the TriGuard™ HDH Embolic Deflection Device During Transcatheter Aortic Valve Implantation
Brief Title: DEFLECT III: A Prospective, Randomized Evaluation of the TriGuard™ HDH Embolic Deflection Device During TAVI
Acronym: TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keystone Heart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEFLECT III
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVR; TAVI; Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- unprotected TAVI (No Intervention): standard unprotected Transcatheter Aortic Valve Implantation
- TAVI with the TriGuard HDH (Experimental): TAVI with the TriGuard HDH embolic deflection device
  Interventions: Device: TriGuard HDH

INTERVENTIONS:
Device: TriGuard HDH — TAVI with the TriGuard HDH embolic deflection device
  Other Names: TriGuard HDH embolic deflection device
  Arms: TAVI with the TriGuard HDH

SUMMARY:
A randomized evaluation of the TriGuard™ HDH embolic deflection device during transcatheter aortic valve implantation.

DETAILED DESCRIPTION:
The TriGuard HDH device is an aortic embolism deflection device intended to reduce the amount of embolic material that may enter the carotid, subclavian, and vertebral arteries during transcatheter heart valve implantation.

To assess the safety, efficacy, and performance of the TriGuard HDH embolic deflection device in patients undergoing transcatheter aortic valve implantation (TAVI), in comparison with patients undergoing unprotected TAVI.

Subjects with indications for TAVI and who meet study eligibility criteria will be randomized 1:1 to one of two treatment arms:

* Intervention - TAVI with the TriGuard HDH embolic deflection device
* Control - standard unprotected TAVI

ELIGIBILITY:
Inclusion Criteria:

* The patient is a male or non-pregnant female ≥18 years of age
* Patient meets indications for TAVI
* The patient is willing to comply with protocol-specified follow-up evaluations
* The patient, or legally authorized representative, has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the appropriate Medical Ethics Committee (EC) or Institutional Review Board (IRB)

Exclusion Criteria:

* Patients undergoing TAVI via the trans-axillary, trans-subclavian, or trans-aortic route
* Patients undergoing TAVI via the transapical approach due to friable or mobile atherosclerotic plaque in the aortic arch
* Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to index procedure per site standard test
* Patients with known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure (according to definition) or AMI >72 hours preceding the index procedure, in whom creatine kinase and creatine kinase-Muscle Brain have not returned to within normal limits at the time of procedure.
* Patients who are currently experiencing clinical symptoms consistent with new-onset AMI, such as nitrate-unresponsive prolonged chest pain
* Patients with a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated, or who will refuse transfusion
* Patients with known other mental or physical illness or known history of substance abuse that may cause non-compliance with the protocol, confound the data interpretation, or is associated with a life expectancy of less than one year
* Patients with severe allergy to heparin or known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel, nitinol, stainless steel alloy, and/or contrast sensitivity that cannot be adequately pre-medicated
* Patients with a history of a stroke or transient ischemic attack (TIA) within the prior 6 months
* Patients with an active peptic ulcer or history of upper gastrointestinal (GI) bleeding within the prior 6 months
* Patients with renal failure (estimated Glomerular Filtration Rate [estimated Glomerular Filtration Rate] <30 mL/min, calculated from serum creatinine by the Cockcroft-Gault formula)
* Patients with hepatic failure (Child-Pugh class C)
* Patients with hypercoagulable states that cannot be corrected by additional periprocedural heparin
* Patients presenting with cardiogenic shock or severe hypotension (systolic blood pressure <90 mm Hg) at the time of the index procedure
* Patients with severe peripheral arterial disease that precludes delivery sheath vascular access
* Patients with a heavily calcified or severely atheromatous aortic arch
* Patients with an innominate artery ostium diameter <11 mm
* Patients with a transverse aortic diameter >40 mm
* Patients with anatomic irregularities of the aortic arch or innominate artery that could prevent positioning and stability of the device
* Patients with contraindication to cerebral MRI
* Patients who have a planned treatment with any other investigational device or procedure during the study period
* Patients planned to undergo any other cardiac surgical or interventional procedure (e.g., concurrent coronary revascularization) during the TAVI procedure or within two (2) weeks prior to the TAVI procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
In hospital procedural safety | Up to 7 days during post procedure hospitalization
  In-hospital procedural safety, defined as the composite of the following Major Adverse Cardiovascular and Cerebrovascular Events (MACCE):
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life threatening (or disabling) bleeding
  * Acute kidney injury - Stage 2 or 3 (including renal replacement therapy)
  * Major vascular complications

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Baumbach, Md., Principal Investigator — Bristol Heart Institute
Locations (14):
- France (3):
  - Hôpital de la Cavale Blanche, Brest
  - Chru-Lille, Lille
  - Clinique chez APHM, Marseille
- Germany (4):
  - Praxisklinik Herz Und Gefässe, Dresden
  - Universitäts-Herzzentrum Freiburg, Freiburg im Breisgau
  - Medical Care Center, Hamburg
  - Städtische Kliniken Neuss, Neuss
- Israel (2):
  - Rambam Medical Center, Haifa
  - Shaarey Tzedek, Jerusalem
- Ferrarotto hospital, Catania, Italy
- UMC Utrecht, Utrecht, Netherlands
- United Kingdom (3):
  - Royal Sussex County Hospital, Brighton
  - Bristol Heart Institute, Bristol
  - Leeds General Infirmary, Leeds